CLINICAL TRIAL: NCT07247123
Title: Protocol for Developing and Testing the Effectiveness of a Skin Cancer Self-Detection Educational Program: A Randomised Controlled Trial
Brief Title: Developing and Testing the Effectiveness of a Skin Cancer Self-Detection Educational Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024/00074
Record Dates: First submitted 2025-11-19; First posted 2025-11-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: Skin Cancer; Skin Cancer Prevention; Benign Skin Growth
Keywords: skin cancer; skin cancer education; skin cancer intervention; patient education; digital education
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Participants will fill up a baseline competency examination and questionnaire, and another at the 4 month mark. Access to the intervention for control group participants will only be provided after the 4-month questionnaire is completed.
  Interventions: Behavioral: Wait-list Control
- Intervention with gain framing (Experimental): Participants will fill up a baseline competency examination and questionnaire. Afterwards, they will have access to a website with gain-framed messages emphasising benefits of adopting a behaviour. Thereafter, another competency questionnaire will be administered following completion of material.
  Interventions: Behavioral: Skin Cancer Self-Detection Educational Program with gain-framing
- Intervention with loss framing (Experimental): Participants will fill up a baseline competency examination and questionnaire. Afterwards, they will have access to a website with loss-framed messages highlighting consequences of failing to adopt a behaviour. Thereafter, another competency questionnaire will be administered following completion of material.
  Interventions: Behavioral: Skin Cancer Self-Detection Educational Program with loss-framing

INTERVENTIONS:
Behavioral: Skin Cancer Self-Detection Educational Program with gain-framing — This educational website will feature gain-framing messages, emphasizing the benefits of adopting a behavior, utilising positive language and analogies. The interventional domains are (1) Education on skin cancer risk factors and epidemiology, (2) UV Protection Advice, (3) Skin Self-Examination Techniques and (4) Differentiating benign vs malignant skin conditions.
  Arms: Intervention with gain framing
Behavioral: Skin Cancer Self-Detection Educational Program with loss-framing — This educational website will feature loss-framing messages, highlight the consequences of failing to adopt a behavior, utilising negative language and analogies. The interventional domains are (1) Education on skin cancer risk factors and epidemiology, (2) UV Protection Advice, (3) Skin Self-Examination Techniques and (4) Differentiating benign vs malignant skin conditions.
  Arms: Intervention with loss framing
Behavioral: Wait-list Control — Participants in the control group will gain access to the intervention websites after the 4-month questionnaire is completed.
  Arms: Control

SUMMARY:
Skin cancer is a significant public health concern, even in an Asian society like Singapore where it ranks among the top 10 cancers. This RCT tests the effectiveness of a skin cancer educational intervention to improve skin cancer outcomes among skin-of-color individuals, including the effects of gain versus loss framing.

DETAILED DESCRIPTION:
Reducing skin cancer related morbidity and mortality involves two broad domains; (1) Identification and early detection of skin cancers and (2) Awareness and behavioral change to reduce modifiable risk factors like UV exposure. Regular self-examination and public education have been shown in RCTs to improve knowledge and identification of skin cancers. However most of these existing studies and the tools they utilise rely on Western-centric photographs and messaging, such as the 'ABCDE rule' for superficial spreading and nodular melanoma. These neglect skin cancers far more common in skin of colour population such as acral lentiginous melanomas, pigmented basal cell and squamous cell carcinomas.

In addition to improving detection, effective behavioural change strategies are needed to encourage protective practices such as regular sunscreen use. Message framing has gained interest as a behavioral change technique: gain-framed messages emphasize the benefits of adopting a behavior, while loss-framed messages highlight the negative consequences of not doing so. Although message framing is widely used in health communication, evidence of its effectiveness in promoting skin cancer-related behaviors is unclear.

Effectiveness of our proposed intervention can help to increase adoption of sun protective behaviours, improve detection rates of skin cancer and allow earlier medical intervention, hence reducing morbidity and mortality of skin cancer.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 16 and above
* Able to read and converse in English
* Able to provide informed consent
* Having the ability to use and interact with a web server or application.

Exclusion Criteria:

- Individuals who have cognitive impairment or decline to participate. There will be no exclusion criteria based on a previous history of skin cancer.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in competency scores | Baseline, immediately post-intervention (for intervention arms), 4 months post-intervention
  Scores measured as percentage of correct questions answered. Range from 0% to 100% with higher score indicating higher ability to differentiate benign from malignant skin lesions.
  Change in scores will be calculated and compared between
  1. Both intervention arms with the control group at 4 months, and
  2. Between gain framed and loss framed intervention arms at 4 months

SECONDARY OUTCOMES:
Knowledge of skin cancer, sun protection and skin self-examination | Baseline, immediately post-intervention (for intervention arms), 4 months post-intervention
  20 Multiple Choice Questions created based on intervention website. Score range from 0 to 20, with a higher score indicate higher knowledge in risks of skin cancer, appropriate sunscreen use and features of cancerous lesions.
Attitudes toward carrying out sun protection behaviours | Baseline, immediately post-intervention (for intervention arms), 4 months post-intervention
  6 questions graded on a 7-point Likert scale, with higher scores indicating better attitudes toward sun protection behaviours
Subjective norms, which refer to participants' perception of whether significant individuals in their lives would support sun protection behaviours | Baseline, immediately post-intervention (for intervention arms), 4 months post-intervention
  7 questions graded on a 7-point Likert scale, with higher scores indicating a greater influence of others' perception on their sun protection behaviours
Behavioural outcomes (sun protection behaviour and skin self-examination) | Baseline, immediately post-intervention (for intervention arms), 4 months post-intervention
  Sun Exposure and Protection Index. 9 questions graded on a 5-point Likert scale assessing sun habits and sun protection behaviour. Lower scores indicate more optimal sun protection behaviours, with an additional adapted question.
  11 additional questions regarding participants' sunscreen usage (e.g. type of sunscreen, frequency of reapplication), and skin-self examination, with a lower score indicating more optimal sun protection behaviours.
Intentions of participants toward carrying out skin cancer risk prevention strategies | Baseline, immediately post-intervention (for intervention arms), 4 months post-intervention
  Sun Exposure and Protection Index (6 questions with an additional adapted question). Each given response score (0-4) are summed, with scores ranging from 0-24, with higher score indicating a low propensity to increase sun protection.
  2 additional questions regarding participants' intentions of conducting a skin-self examination. 7 point Likert Scale (1-7), with higher score indicating higher intentions of conducting a skin-self examination.

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Choi, MBBS, Principal Investigator — National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Yes
IPD shared includes de-identified demographics and measures.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: IPD and supporting information will be available from the time of publication and for four years thereafter.
Access Criteria: Deidentified individual participant data supporting the findings of this study will be available from the corresponding author upon reasonable request. Access will be granted on a case-by-case basis following review and approval of a data access proposal and completion of a data sharing agreement.